CLINICAL TRIAL: NCT01698372
Title: Negative Pressure Dressing to Decrease the Incidence of Leg Wound Complications After CABG
Brief Title: Negative Pressure Dressing After Saphenous Vein Harvest
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: KCI USA, Inc (Industry)
Responsible Party: Principal Investigator, Dr. Paul Fedak, Associate Professor, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: KCI VAC Study
Record Dates: First submitted 2012-09-18; First posted 2012-10-03 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Coronary Artery Disease; Complication of Coronary Artery Bypass Graft; Wound Complication
Keywords: Cardiac surgery.; Wound healing.; Leg wound infection.; Wound care.
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prevena device (Group A) (Experimental): Group A will have the VAC Prevena portable device applied to the saphenous vein harvest site after standard wound closure following coronary artery bypass surgery.
  Interventions: Device: Prevena device (Group A)
- Conventional dressing (Group B) (No Intervention): Group B will have conventional dry dressing applied to the saphenous vein harvest site after standard wound closure following coronary artery bypass surgery.

INTERVENTIONS:
Device: Prevena device (Group A) — This portable device is applied to initiate negative pressure therapy to a wound site.
  Other Names: Prevena Incision Management System; Prevena 125; PRE1001.S Prevena Incision Kit
  Arms: Prevena device (Group A)

SUMMARY:
This study will test the effectiveness of negative pressure wound therapy (using the VAC Prevena device, KCI Canada Inc.) applied to the saphenous vein harvest site after Coronary Artery Bypass Grafting (CABG). When initiated immediately after surgery, this intervention may decrease the incidence of wound infection and non-infectious wound complications. It may decrease wound discomfort and improve mobility and functional recovery of the leg.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting for elective or semi-elective isolated first-time CABG surgery with harvesting of the greater saphenous vein.
* Must be 18 years or older.
* Must live with one hour driving distance from Calgary.
* Must provide written consent.

Exclusion Criteria:

* Previous CABG surgery or previous lower leg surgical intervention.
* In emergent need for surgery.
* Have severe peripheral vascular disease.
* Do not speak and read the English language.
* Have dialysis-dependent renal failure.
* Require chronic steroids.
* Unable to return to clinic for follow-up due to functional or cognitive impairment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2012-09; Primary Completion 2014-11 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline ASEPSIS score of wound healing at 6 weeks. | Baseline and 6 weeks
  The ASEPSIS quantitative wound scoring method will be used to assess patients' leg wound healing after saphenous vein harvesting for coronary artery bypass surgery.

SECONDARY OUTCOMES:
Total score of pain level. | Baseline and 6 weeks
  Patients will be asked to evaluate the level of pain (using the Leg Incision Assessment Form) at the wound site after saphenous vein harvesting.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Fedak, MD, PhD, Principal Investigator — University of Calgary
Locations (1):
- Libin Cardiovascular Institute, Foothills Medical Centre, Calgary, Alberta, Canada

REFERENCES:
- [Derived] Lee AJ, Sheppard CE, Kent WD, Mewhort H, Sikdar KC, Fedak PW. Safety and efficacy of prophylactic negative pressure wound therapy following open saphenous vein harvest in cardiac surgery: a feasibility study. Interact Cardiovasc Thorac Surg. 2017 Mar 1;24(3):324-328. doi: 10.1093/icvts/ivw400. PMID 28025309